CLINICAL TRIAL: NCT04688554
Title: Psychosocial, Behavioral, and Radiologic Changes Following Neurologic Events or Interventions: A Prospective, Non-Interventional, Observational Study
Brief Title: Psychosocial, Behavioral, and Radiologic Changes Following Radiosurgery for Benign Neurologic Disease
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Varian Medical Systems (Industry)
Responsible Party: Principal Investigator, Anthony Cmelak, Professor, Department of Radiation Oncology, Vanderbilt University Medical Center
Other Study IDs: 200209
Record Dates: First submitted 2020-09-16; First posted 2020-12-30 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Obsessive-Compulsive Disorder; Pain, Intractable; Depression
Keywords: Stereotactic Radiosurgery; Cingulotomy; Capsulotomy
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Pain, Intractable; Depression | interventions — Magnetic Resonance Imaging; Diffusion Tensor Imaging; Behavior Rating Scale

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (4):
- Refractory Obsessive Compulsive Disorder: fMRI, DTI, behavioral, psychological, and disease-specific changes following radiosugical capsulotomy
  Interventions: Diagnostic Test: fMRI and DTI; Behavioral: Behavioral questionnaires; Behavioral: Disease-Specific Patient-Reported Outcomes; Behavioral: Behavioral tests
- Refractory Pain: fMRI, DTI, behavioral, psychological, and disease-specific changes following radiosugical cingulotomy
  Interventions: Diagnostic Test: fMRI and DTI; Behavioral: Behavioral questionnaires; Behavioral: Disease-Specific Patient-Reported Outcomes; Behavioral: Behavioral tests
- Refractory Tremor: fMRI, DTI, behavioral, psychological, and disease-specific changes following radiosugical thalamotomy
  Interventions: Diagnostic Test: fMRI and DTI; Behavioral: Behavioral questionnaires; Behavioral: Disease-Specific Patient-Reported Outcomes; Behavioral: Behavioral tests
- Refractory Depression: fMRI, DTI, behavioral, psychological, and disease-specific changes following radiosugical cingulotomy
  Interventions: Diagnostic Test: fMRI and DTI; Behavioral: Behavioral questionnaires; Behavioral: Disease-Specific Patient-Reported Outcomes; Behavioral: Behavioral tests

INTERVENTIONS:
Diagnostic Test: fMRI and DTI — Neurologic imaging correlates
Behavioral: Behavioral questionnaires — RAND 36-item Quality of Life survey, Mini Mental Status Exam, MOCA Cognitive Exam
Behavioral: Disease-Specific Patient-Reported Outcomes — Y-BOCS Survey, QUEST, PDQ39, PHQ2 Depression Screening, PHQ9 Depression Inventory, Beck's Depression Inventory, PROMIS Pain Intensity Short Form 3, McGill Pain Scale, Visual Analog pain scale, FTM (Tremor Scale)
Behavioral: Behavioral tests — Behavioral tests may include one or more of the following procedures: Upper extremity testing, Perdue Peg Board testing, Hand tactile detection and discrimination test, Temperature and pain threshold testing, Lower extremity Testing, Myomotion Inertial Motion Testing.

SUMMARY:
A number of studies from the literature suggest important behavioral, psychosocial, or radiologic changes occur following significant neurologic events or interventions such as stroke, neurosurgery, medications, radiation, systemic therapy, or injury. The purpose of this study is to describe these changes with advanced neurologic imaging and targeted neurologic and neuropsychiatric assessments. This is a non-interventional observational study of minimal risk to participants as there is no medical intervention. The results of this study will be used to inform patients, scientists, and society in the development of future treatments.

DETAILED DESCRIPTION:
Functional magnetic resonance imaging (fMRI) and diffusion tensor tractography (DTI) have rapidly expanded since its emergence two decades ago. fMRI is well established as the single most powerful method for detecting changes in neural activity in vivo, albeit indirectly by detection of changes in blood oxygenation level dependent (BOLD) signals that reflect hemodynamic changes subsequent to neural activity. A conventional fMRI experiment involves the comparison of two or more brain states followed by statistical tests to identify which brain regions were involved in a particular task. The identification of patterns of highly correlated low-frequency MRI signals in the resting brain provides a powerful approach to delineate and describe neural circuits, and an unprecedented ability to assess the manner in which distributed regions work together to achieve specific functions. Since the first reports of temporal correlations in BOLD baseline signals, several distinct cortical long-range networks have been identified and characterized in the resting state, including a default mode network. Moreover, observations of altered resting state connectivity in several disorders and as a function of behavior or cognitive skills suggest these correlations reflect an important level of brain organization and may play a fundamental role in the execution and maintenance of various brain functions. DTI is also an exceedingly important imaging modality that has elucidated the neural connectivity inherent between various cortical and subcortical structures. DTI is routinely used and has enhanced our understanding of functional connections between various parts of the brain. Prior to interventions, DTI is commonly obtained, so that interventionists can avoid critical circuitry. There is suggestion that both fMRI and DTI imaging is influenced by organic or interventional variables, however this is understudied. The neuroscientists and clinicians would greatly value information that would expand our working knowledge of the basic neural substrates and functional neural changes that occur in patients organically or after interventions. A non-invasive, non-interventional, observational study is needed to show the changes that happen to patients organically or in standard of care settings. A greater working understanding of the neural connectivity and changes that happen in the brain is of great future benefit to patients, science, and society as well as future therapeutic development such as post-stroke care, rehabilitation, post-traumatic brain injury, or post-treatment care in the brain that has previously been influenced by intervention or disease.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old and willing and able to sign a written informed consent.
* Eligible for Brain MRI
* History of neurologic event or intervention OR future planned neurologic intervention

Exclusion Criteria:

* Contraindications to MRI of the brain
* Patient declining participation in study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: VUMC adult patients with neurologic disease or patients with neurologic interventions such as neurosurgical procedures or radiation therapy. Men and women of any ethnicity, race or socioeconomic status who meet inclusion criteria will be offered enrollment into the study. Patient will be greater than 18 years of age and meet inclusion and exclusion criteria. Patients eligible for this study will include patients with neurologic events, including but not limited to stroke, depression, infections, psychiatric disease. Intervention is not part of this study, however, patients receiving neurologic interventions, such as neurosurgical procedures or radiation therapy, would be eligible.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2020-08-25 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Describe changes in Obsessive Compulsive Disorder disease burden after stereotactic radiosurgery. | Every 3 months for 1 year or through study completion
  Yale-Brown Obsessive Compulsive Scale questionnaire
Describe changes in Depression disease burden after stereotactic radiosurgery. | Every 3 months for 1 year or through study completion
  Beck's Depression inventory
Describe changes in Pain disease burden after stereotactic radiosurgery. | Every 3 months for 1 year or through study completion
  McGill Pain Scale

SECONDARY OUTCOMES:
Describe changes in cognition after stereotactic radiosurgery. | Every 3 months for 1 year or through study completion
  Montreal Cognitive Assessment
Describe changes in radiologic parameters after stereotactic radiosurgery. | Every 6 months for 1 year or through study completion
  Brain MRI

CONTACTS AND LOCATIONS:
Overall Officials: Anthony J Cmelak, MD, Study Chair — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Research data will be shared upon reasonable request to the principal investigator.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will become available after the publication of the study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-18): https://cdn.clinicaltrials.gov/large-docs/54/NCT04688554/Prot_SAP_000.pdf